CLINICAL TRIAL: NCT01091038
Title: Improving Safety by Basic Computerizing Outpatient Prescribing
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Joseph M Overhage, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 0008-44
Record Dates: First submitted 2010-03-19; First posted 2010-03-23 (Estimated); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Adverse Drug Events
Keywords: Adverse drug events; medical errors; computerized physician order entry; clinical decision support
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine Care (Placebo Comparator): Usual care of patients in the ambulatory setting
  Interventions: Other: Routine Care
- Basic Clinical Decision Support (Experimental): Providers use basic clinical decision support
  Interventions: Other: Basic Clinical Decision Support

INTERVENTIONS:
Other: Basic Clinical Decision Support — The computerized physician order entry (CPOE) intervention provides physicians with a menu of medications from the formulary, default doses, and a range of potential doses for each medication. Physicians were required to enter dosage, route, and frequency for all orders. Also, CPOE ensured that all orders were legible and included the prescribing physician's signature. For a number of medications, the system displayed relevant laboratory results on the screen at the time of ordering. Other features included consequent orders, which are orders that should follow from other orders, and drug-allergy checking, drug-drug interaction checking, and drug-laboratory checking. This included checking for the most frequent drug allergies, about 80 carefully selected drug-drug interactions, and several drug-laboratory combinations
  Arms: Basic Clinical Decision Support
Other: Routine Care — Routine Care
  Arms: Routine Care

SUMMARY:
The study will measure the effect of basic clinical decision support on medical errors and adverse drug events in the ambulatory setting.

ELIGIBILITY:
Inclusion Criteria:

* provider practicing at sites implementing order entry with basic clinical decision support using either the longitudinal medical record (LMR) or Medical Gopher

Exclusion Criteria:

* provider or practice unwilling to participate

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2001-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Adverse Drug Events | 6 months
  Adverse drug events are measured through use of a computerized surveillance system augmented by focused structured human review
Medical Errors | 6 months
  Medical Errors are identified through a computerized surveillance system with structured human review

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Overhage, MD, PhD, Principal Investigator — Indiana University; David Bates, MD, Principal Investigator — Brigham and Women's Hospital; Tejal Gandhi, MD, Principal Investigator — Brigham and Women's Hospital; Andrew Seger, PharmD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Wishard Helath Services, Indianapolis, Indiana
  - Partner's Healthcare, Boston, Massachusetts

REFERENCES:
- [Background] Hope C, Overhage JM, Seger A, Teal E, Mills V, Fiskio J, Gandhi TK, Bates DW, Murray MD. A tiered approach is more cost effective than traditional pharmacist-based review for classifying computer-detected signals as adverse drug events. J Biomed Inform. 2003 Feb-Apr;36(1-2):92-8. doi: 10.1016/s1532-0464(03)00059-5. PMID 14552850